CLINICAL TRIAL: NCT03716583
Title: MELADERM-trial: Melatonin Cream Against Acute Radiation Dermatitis in Patients With Early Breast Cancer: a Pivotal Phase 2, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Melatonin Cream Against Acute Radiation Dermatitis in Patients With Early Breast Cancer
Acronym: MELADERM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dennis Bregner Zetner (Other)
Responsible Party: Sponsor-Investigator, Dennis Bregner Zetner, Principal Investigator, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-001705-91
Record Dates: First submitted 2018-10-16; First posted 2018-10-23 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Radiation Dermatitis; Radiation Dermatitis Acute; Breast Cancer
Keywords: melatonin
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms | interventions — Melatonin; Dimethyl Sulfoxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin/DMSO (Experimental): 25 mg melatonin in 1 g cream twice daily for the duration of the radiation therapy
  Interventions: Drug: Melatonin; Drug: Dimethyl Sulfoxide
- Placebo (Placebo Comparator): 1 g of cream once daily
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Melatonin — 25 mg
  Arms: Melatonin/DMSO
Drug: Dimethyl Sulfoxide — 150 mg
  Arms: Melatonin/DMSO
Drug: Placebos — 1 g
  Arms: Placebo

SUMMARY:
The aim of the present randomized double-blinded placebo-controlled clinical trial is to investigate if melatonin can protect against acute radiation dermatitis in patients with early breast cancer receiving radiation therapy, and whether this has an impact on the patients' quality of life.

DETAILED DESCRIPTION:
The study will be a randomized, placebo-controlled, double-blinded clinical pivotal trial. Patients will be allocated in a ratio of 1:1 to the melatonin or placebo group. Patients will be stratified according to the type of surgery (lumpectomy or mastectomy). Randomization will be performed in blocks of randomized sizes. The study will be performed in the Department of Oncology, Rigshospitalet, Denmark.

Eligible patients with early breast cancer receive adjuvant radiation therapy over 15 to 30 daily fractions (5 fractions per week) of ionizing megavoltage photon radiation to a total of 40 - 60 Gy within 3-5 weeks according to the guidelines of the Danish Breast Cancer Cooperative Group. In this study, the patients will administer approximately 1 g of cream containing melatonin (25 mg/g) and dimethyl sulfoxide (DMSO) (150 mg/g) or a placebo cream topically twice daily on the irradiated skin area. The patients are scheduled to do this every day from the first to the last fraction of radiation therapy, including the days where they do not receive radiation therapy. The investigators have chosen placebo as the comparator due to it being safe and the most reasonable method of evaluating any effects of the intervention. On days where the patients receive radiation, the melatonin/DMSO or placebo cream will be applied no less than 2 hours prior to radiation. Throughout the study, the patients will meet with an investigator once weekly who will monitor compliance and assess outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with early breast cancer
* Over 49 years old
* Have had radical tumor resection surgery
* Follows treatment regimens and follow-up at Rigshospitalet
* Written informed consent after written and verbal information

Exclusion Criteria:

* Inability to understand Danish, written or spoken
* Mental illness (Defined as having a diagnosis and being in medical treatment, or if anticipated poor compliance)
* Previous therapy with ionizing radiation in the thoracic or neck area
* Use of bolus for radiation therapy (A bolus is a material which has dose absorption properties equivalent to tissue. It is placed on the irradiated area to alter dosing or target of the radiation therapy)
* Pregnancy

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Radiation Therapy Oncology Group's acute radiation morbidity scoring criteria of the skin | Once weekly for 8 weeks
  This scale ranges from 0 to 4, being:
  0: No change over baseline
  1. Follicular, faint or dull erythema/epilation/dry desquamation/decreased sweating
  2. Tender or bright erythema, patchy moist desquamation/moderate edema
  3. Confluent, moist desquamation other than skin folds, pitting edema
  4. Ulceration, hemorrhage, necrosis
Erythema evaluated through pixel analysis of clinical photographs | Once weekly for 8 weeks
  Erythema has previously been evaluated by a validated method using software analysis (Image J, version 1.45S, National Institute of health, USA) of digital photos [32]. A "color space converter" function will be used to convert the clinical photos into grayscale in the software analysis. Erythema will be quantified by pixel color analyses where all white colored pixels represent erythema. An a*-value will represent degree of erythema (high a*-values represent a high degree of erythema).
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Breast symptoms (QLQ-BR23) | Once weekly for 8 weeks
  The quality of life questionnaire determines patient-reported quality of life through a series of questions. All questions in the BR23-module (Breast cancer module) are answered on a scale of 1-4, meaning:
  1. Not at all
  2. A little
  3. A lot
  4. Very much The questions vary between symptoms, feelings and activities of daily living.
  Only item 20-23 (specifically questions about the breast area) are defined as a primary outcome. All other outcomes in the questionnaire are considered secondary outcomes.

SECONDARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core module (QLQ-C30) | Once weekly for 8 weeks
  The quality of life questionnaire determines patient-reported quality of life through a series of questions. 28 of 30 questions in the C30-module (Core questionnaire) are answered on a scale of 1-4, meaning:
  1. Not at all
  2. A little
  3. A lot
  4. Very much The questions vary between symptoms, feelings and activities of daily living.
  The remaining two questions are answered on a scale of 1 (Very bad) to 7 (Very well).
European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Breast symptoms (QLQ-BR23) | Once weekly for 8 weeks
  The quality of life questionnaire determines patient-reported quality of life through a series of questions. All questions in the BR23-module (Breast cancer module) are answered on a scale of 1-4, meaning:
  1. Not at all
  2. A little
  3. A lot
  4. Very much The questions vary between symptoms, feelings and activities of daily living.
  Item 1-19 are defined as a secondary outcomes outcome.
Patient reported steroid cream usage | Once weekly for 8 weeks
  Patients will be questioned once weekly about usage of steroid cream. The questions will be:
  Have you used any steroid cream throughout your radiation therapy? (Yes/No) If yes, when did you begin using steroid cream? (Date) If yes, how many days have you used steroid cream? (Number of days)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis B Zetner, MD, Principal Investigator — Center for Perioperativ Optimization
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT03716583/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT03716583/ICF_001.pdf